CLINICAL TRIAL: NCT06107439
Title: Impact of Lipodystrophy on the Inflammatory State of Non-diabetic Dunnigan Reunion Island Subjects
Acronym: LIPOKINES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021/CHU/12
Record Dates: First submitted 2023-09-14; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: Lipodystrophy; Dunnigan Syndrome
MeSH Terms: conditions — Lipodystrophy; Lipodystrophy, Familial Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sampling and clinical data collection (Other): Participant blood and urine are sampled for inflammatory signal analysis
  Interventions: Biological: Bood and urine sampling

INTERVENTIONS:
Biological: Bood and urine sampling — Bood and urine sampling

SUMMARY:
Few data and small numbers affect the inflammatory profile of Dunnigan patients. The levels of certain pro-inflammatory biomarkers would be found higher in these subjects compared to control individuals. However, in these studies, several confounding factors were not taken into account such as smoking, an underlying chronic inflammatory disease such as diabetes and could limit the interpretation of the results. There is no other observation of the anti-inflammatory status of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (>18 years old) affected by partial Dunnigan lipodystrophy in the homozygous or heterozygous state (genetic search for the positive mutation carried out before inclusion in the study).
* Person affiliated to or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator.

Exclusion Criteria:

* - Minor
* Persons placed under judicial protection, person participating in another research including a period of exclusion still in progress, severely impaired physical and/or psychological health, which, according to the investigator, may affect the participant's compliance with the study
* Previous known diabetes
* Pregnant woman
* Woman who gave birth less than 6 months ago
* Breastfeeding in progress
* Participation in other research that may have an impact on the evaluation of the main judgment criteria
* Hemoglobin b level < 7 mg/dl or < 9-10 mg/dl for patients with cardiovascular or respiratory pathology.
* Proven inflammatory pathologies
* Anti-inflammatory treatment: taking corticosteroids in the last 3 months.
* Active smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2025-08-13 (Estimated)

PRIMARY OUTCOMES:
pro-inflammatory markers | inclusion day
  blood sample and dosage of pro inflammatory cytokine

CONTACTS AND LOCATIONS:
Locations (1):
- CHU La Réunion DRCI, Saint-Pierre, Reunion